CLINICAL TRIAL: NCT01799395
Title: Prevalence, Incidence and Predictors of Central Airway Obstruction in Patients With Advanced Lung Cancer
Brief Title: Prevalence and Incidence of Central Airway Obstruction in Advanced Lung Cancer
Status: Terminated | Type: Observational
Why Stopped: Staff constraints made it impossibile to enroll consecutive patients, making the sample not representative of the true cancer population
Sponsor: Maggiore Bellaria Hospital, Bologna (Other)
Responsible Party: Principal Investigator, Rocco Trisolini, M.D., Maggiore Bellaria Hospital, Bologna
Other Study IDs: 13002-Trisolini
Record Dates: First submitted 2013-02-23; First posted 2013-02-26 (Estimated); Last update posted 2017-09-12 (Actual); Status verified 2017-09

CONDITIONS: Lung Cancer
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Lung Cancer: All patients with advanced lung cancer candidate for chemotherapy or chemotherapy + radiation therapy will be enrolled and followed-up for 1 year clinically and radiologically (Chest CT) to verify whether or not central airway obstruction is present at the time of diagnosis or occurs in the year following diagnosis (or in the life span from diagnosis and death in patients who die before 1 year of diagnosis). Furthermore, predictor variables possibly associated with central airway obstruction will be studied.

SUMMARY:
Lung cancer may cause central airway obstruction through several different mechanisms (invasion by the primary tumor, invasion by metastatic lymph nodes, airway metastasis).

The aim of the present study is to determine the prevalence at the time of diagnosis, the incidence at 1 year from the diagnosis, and the predictors of central airway obstruction associated with advanced lung cancer.

ELIGIBILITY:
Inclusion Criteria:

* Advanced lung cancer with indication for chemotherapy or chemotherapy + radiation therapy

Exclusion Criteria:

* Age < 18 year
* Pregnancy
* Refusal to sign informed consent

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with advanced lung cancer undergoing treatment and follow-up at the Oncology Units of the Azienda USL di Bologna (government structure that manages several public hospitals that "cover" a 800.000 inhabitants area)
Sampling Method: Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2013-02; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Incidence of central airway obstruction | 12 months
  The incidence will be measured over a 12 month period after diagnosis (or over the life span from diagnosis to death in patients who die before 1 year from the diagnosis)

SECONDARY OUTCOMES:
Predictor variables associated with the presence/occurrence of central airway obstruction | 12 months
Prevalence of central airway obstruction | 1 day
  The prevalence of central airway obstruction will be evaluated at the time of diagnosis

CONTACTS AND LOCATIONS:
Overall Officials: Rocco Trisolini, M.D., Principal Investigator — Maggiore Bellaria Hospital, Bologna, Italy
Locations (5):
- Italy (5):
  - Bentivoglio Hospital, Bentivoglio, Emilia-Romagna
  - Bellaria Hospital, Bologna, Emilia-Romagna
  - Maggiore Hospital, Bologna, Emilia-Romagna
  - Budrio Hospital, Budrio, Emilia-Romagna
  - SS Salvatore Hospital, San Giovanni in Persiceto, Emilia-Romagna